CLINICAL TRIAL: NCT03561675
Title: Acetazolamide for Prevention of Acute Mountain Sickness in Healthy Lowlanders Older Than 40 Years. Randomized Trial.
Brief Title: Effect of Acetazolamide on Acute Mountain Sickness in Lowlanders Older Than 40 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-01-8/305
Record Dates: First submitted 2018-05-14; First posted 2018-06-19 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Acute Mountain Sickness
Keywords: healthy participants older than 40 years; altitude; prevention; acetazolamide
MeSH Terms: conditions — Altitude Sickness | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 375mg/day (capsule @125 mg: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3'100m until the morning after the second night at 3'100m
  Interventions: Drug: ACETAZOLAMIDE oral capsule
- PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3'100m until the morning after the second night at 3'100m.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ACETAZOLAMIDE oral capsule — Administration of 1x125mg acetazolamide in the morning, 2x125mg in the evening, starting 24 hours before departure to 3'100m
  Arms: ACETAZOLAMIDE oral capsule
Drug: Placebo oral capsule — Administration of equally looking placebo capsules in the morning and evening, starting 24 hours before departure to 3'100m
  Arms: PLACEBO oral capsule

SUMMARY:
Randomized, placebo controlled trial evaluating efficacy of acetazolamide in preventing acute mountain sickness in lowlanders older than 40 years travelling from 760 m to 3'100 m.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the efficacy of acetazolamide prophylaxis in reducing the incidence of acute mountain sickness (AMS) in lowlanders older than 40 years travelling to altitude. Participants living in the Bishkek area, Kyrgyzstan (760m), will be transferred by car within 4h to the Tuja Ashu high altitude clinic (3'100 m), and stay there for 2 days. Acetazolamide 375mg/day (or placebo), will be administered before departure at 760 m and during the stay at altitude. Outcomes will be assessed during the stay at 3'100 m.

An interim analysis will be carried out when 80 participants will have completed the study or after the first year. The Peto's method will be used and the trial will be stopped when pre-specified futility boundaries were crossed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, age 40-75 yrs, without any disease and need of medication.
* Born, raised and currently living at low altitude (<800m).
* Written informed consent.
* Kyrgyz ethnicity

Exclusion Criteria:

* Any active respiratory, cardiovascular or other disease requiring regular treatment or being otherwise relevant for tolerance of hypoxia or altitude exposure.
* Any condition that may interfere with protocol compliance including current heavy smoking (>20 cigarettes per day or >20 pack-years with active smoking during the last 10 years), regular use of alcohol.
* Allergy to acetazolamide and other sulfonamides.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Acute mountain sickness (AMS), incidence | Day 1 to 3 at 3'100m
  Difference between acetazolamide and placebo group in the incidence of AMS during the stay at 3'100 m.

SECONDARY OUTCOMES:
Acute mountain sickness (AMS), severity assessed by the Lake Louise score | Day 1 to 3 at 3'100m
  Difference between acetazolamide and placebo group in the severity of AMS during the stay at 3'100 m. The severity of acute mountain sickness (AMS) will be assessed by the Lake Louise questionnaire (LLS), a validated questionnaire about AMS. The severity will be calculated when the presence of headache and at least one of the following symptoms is present: gastrointestinal upset, fatigue or weakness, dizziness or lightheadedness and difficulty sleeping. Each of the five questions is asked with the corresponding 0 to 3 rating of the response (0 = Not present, 1 = mild, 2 = moderate, 3 = severe). The sum of the responses on these questions is then calculated, resulting in the AMS severity.
Acute mountain sickness (AMS) at 760 m with and without acetazolamide, severity | Day 3 at 760 m
  Difference between acetazolamide and placebo group in the severity of AMS at 760 m.
Altitude related adverse health effects (ARAHE), incidence | Day 1 to 3 at 3'100m
  Difference between acetazolamide and placebo group in the incidence of ARAHE during the stay at 3'100 m.
  ARAHE are defined as the following:
  * Moderate to severe AMS (Lake Louise score ≥3 and/or Environmental Symptoms questionnaire AMSc score ≥0.7) and/or any of the following:
  * Severe hypoxemia (SpO2 at rest <80% for >30 min or <75% for >15 min, exercise oxygen desaturation SpO2 <75% for >1 min accompanied by symptoms or signs of hypoxemia)
  * Symptomatic cardiovascular disease (arterial blood pressure systolic >200 mmHg, diastolic >110 mmHg not responding to blood pressure lowering drugs within 1 hr; chest pain with ECG signs of ischemia or new onset arrhythmia)
  * Withdrawal from the study by the decision of the independent physician for safety reasons or by the patient.
Spirometric measurement of forced expiratory volume in one second | Day 2 at 760m and day 2 at 3'100m
  Difference in altitude-induced change in the forced expiratory volume in one second between the acetazolamide and placebo group
Arterial partical pressure of oxygen | Day 2 at 760m and day 2 at 3'100m
  Difference in altitude-induced changes in arterial partical pressure of oxygen between the acetazolamide and placebo group
Drug side effects | Day 1 to 3 at 3'100m
  Difference between acetazolamide and placebo group in the incidence of medication side effects during the stay at 3'100 m.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan; Michael Furian, MSc, Principal Investigator — University Hospital, Zürich
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

REFERENCES:
- [Derived] Furian M, Mademilov M, Buergin A, Scheiwiller PM, Mayer L, Schneider S, Emilov B, Lichtblau M, Bitos K, Muralt L, Groth A, Reiser AE, Sevik A, Sheraliev U, Marazhapov NH, Aydaralieva S, Muratbekova A, Tabyshova A, Abdraeva A, Buenzli S, Sooronbaev TM, Ulrich S, Bloch KE. Acetazolamide to Prevent Adverse Altitude Effects in COPD and Healthy Adults. NEJM Evid. 2022 Jan;1(1):EVIDoa2100006. doi: 10.1056/EVIDoa2100006. Epub 2021 Dec 22. PMID 38296630
- [Derived] Graf LC, Furian M, Bitos K, Mademilov M, Abdraeva A, Buenzli J, Buenzli S, Aidaralieva S, Sheraliev U, Mayer LC, Schneider SR, Sooronbaev TM, Ulrich S, Bloch KE. Effect of altitude and acetazolamide on sleep and nocturnal breathing in healthy lowlanders 40 y of age or older. Data from a randomized trial. Sleep. 2023 Apr 12;46(4):zsac269. doi: 10.1093/sleep/zsac269. PMID 36356042